CLINICAL TRIAL: NCT06331806
Title: Myocardial Fibrosis Identification in Patients With Anthracycline-induced Cardiotoxicity: Clinical and Prognostic Implications
Brief Title: Myocardial Fibrosis Identification in Patients With Anthracycline-induced Cardiotoxicity
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: European Institute of Oncology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IEO 398
Record Dates: First submitted 2024-03-18; First posted 2024-03-26 (Actual); Last update posted 2024-06-24 (Actual); Status verified 2024-03

CONDITIONS: Cardiomyopathy Due to Drug

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Evaluation of myocardial fibrosis (Other): Echocardiogram with left ventricular ejection fraction (LVEF) evaluation (biplane method) and CMR with contrast media agent
  Interventions: Diagnostic Test: Evaluation of myocardial fibrosis

INTERVENTIONS:
Diagnostic Test: Evaluation of myocardial fibrosis — echocardiogram with left ventricular ejection fraction (LVEF) evaluation (biplane method) and CMR with contrast media agent

SUMMARY:
This is an interventional study for patients who had developed Anthracycline-Induced Cardiotoxicity (AIC) during or after anthracycline-containing therapy, referred to the Cardioncology Unit for heart failure treatment

DETAILED DESCRIPTION:
The main aim of this interventional study is to evaluate biochemical and imaging markers of fibrosis in patients who had previously developed AIC during or after anthracycline-containing therapy.

Anthracycline-induced cardiomyopathy (AIC) is define as a reduction in Left Ventricular Ejection Fraction (LVEF) >10% units from baseline and below 50%, assessed by echocardiography, during or after anthracycline-containing therapy.

All patients will undergo:

* at time 0

  * an echocardiogram with LVEF evaluation (biplane method)
  * a single blood sample.
* at time 1 - a Cardiac Magnetic Resonance (RMC) with contrast agent (T1 mapping technique) (time 1 = within 72 hours from blood sample).

ELIGIBILITY:
Inclusion Criteria:

* Patients who developed AIC during or after anthracycline-containing therapy assessed by LVEF valuation by echocardiography.

Exclusion Criteria:

* Age <18 years
* Contraindications to contrast medium magnetic resonance imaging

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-02-22 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Evaluation of blood levels of Suppression Of Tumorigenicity 2 (ST2) | 1 month
  Evaluation of blood levels of Suppression Of Tumorigenicity 2 (ST2) gene as biomarker of fibrosis
Evaluation of blood levels of Galectin-3 (Gal-3) | 1 month
  Evaluation of blood levels of Galectin-3 (Gal-3) as biomarker of fibrosis
Evaluation of Enhanced Liver Fibrosis score (ELF) | 1 month
  Evaluation of Enhanced Liver Fibrosis score (ELF) as biomarker of fibrosis ELF score is a "marker set" constituted by 3 markers of fibrosis: lhyaluronic acid, amino-terminal propeptide of type III procollagen, and tissue inhibitor of metalloproteinase 1, firstly utilized in the diagnosis and assessment of the severity of liver
Evaluation of CMR imaging marker of fibrosis | 1 month
  Evaluation at CMR of Myocardial T1 before and after contrast media infusion and Myocardial extracellular volume

SECONDARY OUTCOMES:
Evaluation of improvement in left ventricular ejection fraction (LVEF) absolute points from baseline | 1 month
  evaluation of the response to heart failure treatment in terms of improvement in left ventricular ejection fraction (LVEF) absolute points from baseline
Evaluation of levels of Troponin I (TnI) and B-type Natriuretic Peptide (BNP) | 1 month
  Troponin I (TnI) and B-type Natriuretic Peptide (BNP) are biomarkers already utilized in the early diagnosis and monitoring of AIC and recognized prognostic indexes in patients with heart failure.
Evaluation of levels of cytochrome C | 1 months
  cytochrome C is a marker of mitochondrial dysfunction

CONTACTS AND LOCATIONS:
Overall Officials: Daniela Cardinale, MD, Principal Investigator — European Institute of Oncology
Locations (1):
- European Institute of Oncology, Milan, Italy